CLINICAL TRIAL: NCT02155621
Title: Personalized OncoGenomics (POG) Program of British Columbia: Connecting Cancer Genomics to Cancer Care
Brief Title: Personalized Oncogenomics (POG) Program of British Columbia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: POG 4.0
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Cancers; Advanced Cancers; Cancers That Cannot be Treated With Curative Intent
Keywords: cancer genomics; precision medicine; metastatic cancer; clinical decision-making
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genome Sequencing (Experimental): There is only one arm to this study.
  Interventions: Genetic: Genome sequencing

INTERVENTIONS:
Genetic: Genome sequencing — Subjects will have their cancers biopsied and blood samples taken; both will undergo genomic sequencing and analysis

SUMMARY:
The genomic heterogeneity of cancers implies that to effectively use targeted therapies the investigators will need to assess each individual cancer and match it to a biologically relevant targeted therapy. The investigators will use full genome sequencing to try to identify cancer "drivers" and corresponding drugs that may inhibit these pathways.

DETAILED DESCRIPTION:
Carcinogenesis is an immensely complex process such that even within a histologic cancer subtype - for example adenocarcinoma of the lung or breast - there is significant variability in cancer behaviour and response to therapy. Analyses of individual patients demonstrate unique molecular signatures for every cancer examined. Frequently, multiple different pathways are involved in disease growth and progression and the dominant process varies from person to person and perhaps even within different sites of disease within one person. As well these variations evolve in response to treatment.

Recognizing genetic aberrations that promote disease facilitates targeted treatment; this has been demonstrated in several small subgroups of cancers in which specific genetic mutations or translocations have been successfully treated with targeted chemotherapy agents. With many recognized mutations and aberrations, personalized evaluation of the genetic signature encoded in DNA and RNA may provide important diagnostic information and potentially enable directed therapy to the appropriate oncologic pathway thereby providing information to help guide chemotherapy choices

Our initial pilot project demonstrated the feasibility of this approach at our institution (with 100 patients). We now know it is possible to identify and consent patients, sequence the genome and transcriptome, analyze and report abnormalities, and identify potential actionable targets in a clinically relevant time frame.

The Personalized OncoGenomics (POG) program has been operational across the province of BC since 2012. The initial two-year phase established the infrastructure and workflow by which patients with metastatic or incurable cancers could be identified, consented, and biopsied for genomic sequencing in a clinically accredited lab (Laskin et al., 2015). The next phase of the POG program (2014 - 2017) included a strong educational and engagement process such that 83 (80%) of the medical oncologists at BC Cancer were trained to consent and enroll patients onto POG. This means that the oncology community in BC has a broad education in cancer genomics and how these data may be applied to individual patients. Since 2017, the program has been integrated into the Vancouver Cancer Centre's phase 1 clinical trials unit and the focus has shifted to use the study patients and data to address more focused clinical therapeutic trials such as the CCTG CAPTUR study (Skamene et al., 2018). POG-like WGTA has been the driving force behind the creation of the Terry Fox Marathon of Hope Cancer Centre Network (MOHCCN) which is a national program for cancer genomic data sharing across Canada.

The overarching theme of this POG Program is to create a comprehensive cataloguing of somatic cancer mutations and cellular pathway abnormalities that could generate profound insights into genetic patterns that underlie particular cancer phenotypes, and provide valuable prognostic and predictive information.

Eligible subjects will have several samples analyzed: a fresh tumour biopsy (typically 5 cores are required), a blood sample for normal comparison and archival tumours when available. Also, technology has improved such that we may consider using paraffin embedded materials. Comprehensive DNA and RNA sequencing is performed followed by an in-depth bioinformatic analysis to identify somatic mutations, gene expression changes or other abnormalities that might be cancer "drivers" or provide actionable (diagnostic) or druggable targets. The POG team meets every week to discuss the detailed genomic reports for patients, consider additional validation tests when necessary, and debate research questions. The clinicians (typically 5 - 10) come to a consensus on what systemic therapies might be appropriate based on these results. Whenever possible subjects are matched to clinical trials.

ELIGIBILITY:
Inclusion criteria:

1. Patients must agree to allow their archival specimens to be used and possibly completely depleted for these analyses.
2. Willing and able to have a study-specific biopsy or resection of the tumour or metastatic site OR if there is adequate archival material available, either fresh frozen or FFPE (if specimen is thought to be adequate) that is taken after the most recent chemo or radiation. Ideally this sample should have been collected within 16 weeks of the date of consent. If archival tissue is not adequate and if a biopsy is not feasible or deemed medically safe by the investigators the patient would become ineligible.
3. Patients must understand and agree to provide a blood test (or other sample of normal DNA) for germline genomic analysis.
4. ECOG PS 0 or 1.
5. Age >/= 18 years.
6. Estimated life expectancy >/= 6 months and high likelihood of being clinically fit for a therapeutic clinical trial in 3-6 months.
7. Measurable disease with RECIST v1.1 (or updated version).
8. Adequate organ function.
9. Patients must clearly understand that this data may be used to help guide treatment recommendations, including the avoidance of some therapeutic agents or the suggestion to use standard cytotoxic chemotherapy agents.
10. Willingness to have their de-identified genomic and clinical data shared with national and international research collaborators and data sharing platforms (as detailed in the consent form).
11. Willingness to be contacted for future studies based on the data that is generated by participation in POG; included in this is the anticipation that patient would be fit or a candidate for clinical trials.

Exclusion criteria:

1. Unable or unwilling to consent to the above tissue and blood requirements.
2. Significant medical condition that in the opinion of the treating or consenting oncologist and/or the POG central office review team renders the subject not suitable for participation. This includes the likelihood that a subject would be suitable for a clinical trial within 12 weeks after POG biopsy.
3. Unwilling or unable to provide treatment and outcome follow up information to the BC Cancer or affiliated investigators.
4. Unwilling to receive medically actionable findings (germline and/or somatic).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2014-07; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Influence of genomic data on clinical decision-making | 5 years
  This outcome will allow us to study how often in-depth genomic data impacts on clinical decision-making in a general oncology population. It will help describe how useful or important this sort of data is in daily practice.
Cataloging of cancer genomes | 5 years
  Accumulation of genomic information linked to treatment/outcome data will greatly enhance our knowledge and understanding of cancers and response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janessa J Laskin, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Jamshidi F, Pleasance E, Li Y, Shen Y, Kasaian K, Corbett R, Eirew P, Lum A, Pandoh P, Zhao Y, Schein JE, Moore RA, Rassekh R, Huntsman DG, Knowling M, Lim H, Renouf DJ, Jones SJ, Marra MA, Nielsen TO, Laskin J, Yip S. Diagnostic value of next-generation sequencing in an unusual sphenoid tumor. Oncologist. 2014 Jun;19(6):623-30. doi: 10.1634/theoncologist.2013-0390. Epub 2014 May 7. PMID 24807916
- [Background] Jones SJ, Laskin J, Li YY, Griffith OL, An J, Bilenky M, Butterfield YS, Cezard T, Chuah E, Corbett R, Fejes AP, Griffith M, Yee J, Martin M, Mayo M, Melnyk N, Morin RD, Pugh TJ, Severson T, Shah SP, Sutcliffe M, Tam A, Terry J, Thiessen N, Thomson T, Varhol R, Zeng T, Zhao Y, Moore RA, Huntsman DG, Birol I, Hirst M, Holt RA, Marra MA. Evolution of an adenocarcinoma in response to selection by targeted kinase inhibitors. Genome Biol. 2010;11(8):R82. doi: 10.1186/gb-2010-11-8-r82. Epub 2010 Aug 9. PMID 20696054
- [Background] Laskin J, Jones S, Aparicio S, Chia S, Ch'ng C, Deyell R, Eirew P, Fok A, Gelmon K, Ho C, Huntsman D, Jones M, Kasaian K, Karsan A, Leelakumari S, Li Y, Lim H, Ma Y, Mar C, Martin M, Moore R, Mungall A, Mungall K, Pleasance E, Rassekh SR, Renouf D, Shen Y, Schein J, Schrader K, Sun S, Tinker A, Zhao E, Yip S, Marra MA. Lessons learned from the application of whole-genome analysis to the treatment of patients with advanced cancers. Cold Spring Harb Mol Case Stud. 2015 Oct;1(1):a000570. doi: 10.1101/mcs.a000570. PMID 27148575
- [Background] Skamene T, Siu LL, Renouf DJ, Laskin JJ, Bedard PL, Jones SJM, Ferrario C, Whitlock J, Petrie J, Sullivan P, Malone ER, Nomikos D, Chen BE, Dancey Y. Canadian profiling and targeted agent utilization trial (CAPTUR/PM.1): A phase II basket precision medicine trial. J Clin Oncol. 2018;36(15), TPS12127. doi:10.1200/JCO.2018.36.15_suppl.TPS12127
- [Derived] Yu IS, Wee K, Williamson L, Titmuss E, An J, Naderi-Azad S, Metcalf C, Yip S, Horst B, Jones SJM, Paton K, Nelson BH, Marra M, Laskin JJ, Savage KJ. Exceptional response to combination ipilimumab and nivolumab in metastatic uveal melanoma: Insights from genomic analysis. Melanoma Res. 2022 Aug 1;32(4):278-285. doi: 10.1097/CMR.0000000000000810. Epub 2022 Jun 17. PMID 35726793
- [Derived] Lavoie JM, Mitchell T, Lee SE, Deol B, Chia SK, Gelmon KA, Kollmannsberger CK, Tinker AV, Jones SJM, Marra M, Laskin J, Renouf DJ. Patient selection for a developmental therapeutics program using whole genome and Transcriptome analysis. Invest New Drugs. 2020 Oct;38(5):1601-1604. doi: 10.1007/s10637-020-00892-8. Epub 2020 Jan 6. PMID 31907737
- [Derived] Karasinska JM, Topham JT, Kalloger SE, Jang GH, Denroche RE, Culibrk L, Williamson LM, Wong HL, Lee MKC, O'Kane GM, Moore RA, Mungall AJ, Moore MJ, Warren C, Metcalfe A, Notta F, Knox JJ, Gallinger S, Laskin J, Marra MA, Jones SJM, Renouf DJ, Schaeffer DF. Altered Gene Expression along the Glycolysis-Cholesterol Synthesis Axis Is Associated with Outcome in Pancreatic Cancer. Clin Cancer Res. 2020 Jan 1;26(1):135-146. doi: 10.1158/1078-0432.CCR-19-1543. Epub 2019 Sep 3. PMID 31481506
- [Derived] Wong D, Shen Y, Levine AB, Pleasance E, Jones M, Mungall K, Thiessen B, Toyota B, Laskin J, Jones SJM, Marra MA, Yip S. The pivotal role of sampling recurrent tumors in the precision care of patients with tumors of the central nervous system. Cold Spring Harb Mol Case Stud. 2019 Aug 1;5(4):a004143. doi: 10.1101/mcs.a004143. Print 2019 Aug. PMID 31371350
- [Derived] Williamson LM, Steel M, Grewal JK, Thibodeau ML, Zhao EY, Loree JM, Yang KC, Gorski SM, Mungall AJ, Mungall KL, Moore RA, Marra MA, Laskin J, Renouf DJ, Schaeffer DF, Jones SJM. Genomic characterization of a well-differentiated grade 3 pancreatic neuroendocrine tumor. Cold Spring Harb Mol Case Stud. 2019 Jun 3;5(3):a003814. doi: 10.1101/mcs.a003814. Print 2019 Jun. PMID 31160355
- [Derived] Thibodeau ML, Zhao EY, Reisle C, Ch'ng C, Wong HL, Shen Y, Jones MR, Lim HJ, Young S, Cremin C, Pleasance E, Zhang W, Holt R, Eirew P, Karasinska J, Kalloger SE, Taylor G, Majounie E, Bonakdar M, Zong Z, Bleile D, Chiu R, Birol I, Gelmon K, Lohrisch C, Mungall KL, Mungall AJ, Moore R, Ma YP, Fok A, Yip S, Karsan A, Huntsman D, Schaeffer DF, Laskin J, Marra MA, Renouf DJ, Jones SJM, Schrader KA. Base excision repair deficiency signatures implicate germline and somatic MUTYH aberrations in pancreatic ductal adenocarcinoma and breast cancer oncogenesis. Cold Spring Harb Mol Case Stud. 2019 Apr 1;5(2):a003681. doi: 10.1101/mcs.a003681. Print 2019 Apr. PMID 30833417
- [Derived] Wong HL, Yang KC, Shen Y, Zhao EY, Loree JM, Kennecke HF, Kalloger SE, Karasinska JM, Lim HJ, Mungall AJ, Feng X, Davies JM, Schrader K, Zhou C, Karsan A, Jones SJM, Laskin J, Marra MA, Schaeffer DF, Gorski SM, Renouf DJ. Molecular characterization of metastatic pancreatic neuroendocrine tumors (PNETs) using whole-genome and transcriptome sequencing. Cold Spring Harb Mol Case Stud. 2018 Feb 1;4(1):a002329. doi: 10.1101/mcs.a002329. Print 2018 Feb. PMID 29092957
- [Derived] Jones MR, Lim H, Shen Y, Pleasance E, Ch'ng C, Reisle C, Leelakumari S, Zhao C, Yip S, Ho J, Zhong E, Ng T, Ionescu D, Schaeffer DF, Mungall AJ, Mungall KL, Zhao Y, Moore RA, Ma Y, Chia S, Ho C, Renouf DJ, Gelmon K, Jones SJM, Marra MA, Laskin J. Successful targeting of the NRG1 pathway indicates novel treatment strategy for metastatic cancer. Ann Oncol. 2017 Dec 1;28(12):3092-3097. doi: 10.1093/annonc/mdx523. PMID 28950338